CLINICAL TRIAL: NCT03022812
Title: Is E-health a Way to Increase Ability and Health and Make Health Care More Effective in Chronic Whiplash? A Prospective Randomized Controlled Multicenter Trial
Brief Title: Neck-specific Exercise in Chronic Whiplash
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Anneli Peolsson, Professor, PhD, PT, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016/135-31
Record Dates: First submitted 2016-12-20; First posted 2017-01-18 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Whiplash Associated Disorders
Keywords: Neck pain; Rehabilitation; Exercise Therapy; Internet
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercises at a physiotherapy clinic (Active Comparator): Neck-specific exercise at a physiotherapy clinic, 24 times during 12 weeks (plus an additional first visit).
  Interventions: Other: Neck-specific exercise
- Exercises with Internet support (Experimental): Neck-specific exercise with Internet support combined with 3 visits at a physiotherapy clinic (plus an additional first visit), exercises mainly performed outside the health care system during 12 weeks.
  Interventions: Other: Neck-specific exercise

INTERVENTIONS:
Other: Neck-specific exercise — Neck-specific exercise

SUMMARY:
Neck pain is fourth among the most common conditions worldwide associated with longer periods of living with disability. Annually, about 30 000 people in Sweden undergo a whiplash trauma (WAD), and half of those individuals will develop chronic problems with high costs for the individual and society. Evidence for chronic WAD treatment is scarce, although neck-specific training at a physiotherapy clinic (2 times a week for 3 months) has demonstrated good results. A more efficient, flexible rehabilitation with reduced waiting times and lower costs is needed, ideally replacing lengthy on-site treatment series by health care providers. Internet-based care has proven to be a viable alternative to personal care meetings for a variety of diseases and interventions, but studies are lacking on Internet-based interventions for individuals with chronic neck problems. The purpose of this study is to investigate if A) neck-specific training delivered through Internet-based care differs from B) a longer series of treatments at a physiotherapy clinic regarding, e.g., work ability, sick-leave and disability. This prospective, randomized study involves 140 participants. Measurement is done at baseline, 3 months (end of treatment), and 15 months (12 months after end of treatment in the study) and will include ratings of work ability, sick-leave, work presenteeism, disability, pain, health, satisfaction with care, quality of life, and cost-effectiveness. The study results may contribute to the development of a more effective rehabilitation, flexible and equal care, shorter waiting times, increased availability and lower costs for health care and society. The program can be implemented on a broader scale in neck pain patients.

DETAILED DESCRIPTION:
The purpose of the study is to investigate if the effect of neck-specific exercises in people with chronic WAD (at risk for or at sick-leave) differs based on distribution via Internet-based care in combination with three visits (+ a first examination visit due to Swedish law) to the physiotherapist compared to a longer series (2 times/week for 3 months, i.e., 24 times + a first visit) of exercises at the physiotherapy clinic. Outcomes are for instance work ability, sick-leave, physical and psychological disability, pain, quality of life, satisfaction with treatment, and cost effectiveness. Further objectives are to a) describe the level of work ability, work presenteeism, and sick leave; b) determine which factors are related to a good work ability; c) identify factors predictive of a favourable outcome regarding work ability, disability, and pain; and d) describe how the participants perceived an Internet-based rehabilitation.

Hypothesis: Internet-based support combined with a few (three) physiotherapist visits has an equivalent effect to a longer exercise period (24 times) at a physiotherapist clinic and yields lower economic costs for society.

Design This is an experimental, longitudinal, prospective, multicentre randomized controlled trial (RCT) with two treatment arms. Treatment that has previously been shown to be effective (neck-specific exercises guided by a physiotherapist and performed at the physiotherapist clinic) for the current population constitutes the control treatment for the new Internet-based neck-specific exercise treatment. A total of 140 people are expected to be included, 70 in each group (sample size estimated by statisticians). Independent physiotherapists in primary care clinical practice will distribute the treatment. The project manager will not be a test leader.

Recruitment and randomization Interested patients will contact the research team (experienced physiotherapists), and after a small survey filled in by the potential participant, a project team member will perform a telephone interview, ask about the medical history, and perform a physical examination to ensure that criteria for study participation are met. If the study criteria are met and after written and oral informed consent of the patient, the patient will fill out a questionnaire (baseline data) and undergo physical measurements of neck-related function. Baseline measurements must be completed for inclusion.

The patient will be randomized through a computerized randomization list (block randomization conducted by a statistician, stratification by gender) to one of two groups of 3 months of treatment with neck-specific exercises: A) exercises at a physiotherapy clinic 2 times/week for 3 months; or B) Internet-based support exercises in combination with four visits to the physiotherapist. The test leader is blinded for group allocation. The randomization is performed by an independent researcher not otherwise involved in any of the test or treatments. The researcher sends an opaque envelope containing the name and contact details of the patient and information about the randomization group to the treating physiotherapist, who calls the patient to a new clinical examination (by law) before treatment can start. Due to the nature of the study neither participants nor treating therapists can be blinded, however all tests are done by blinded test leaders. Data collection in the form of questionnaires and tests of physical neck-related function occurs at baseline (before randomization) and after 3 months (when the treatment ends) and 15 months (12 months after completion of the intervention in the project). The treating physiotherapists will receive oral and written information and a day of practical training. The treating physiotherapist is also able to consult with the project managers at any time if necessary. An exercise diary is maintained by patients in both groups, and the number of care contacts is recorded by the physiotherapist. Seventy people per group, i.e., a total of 140 participants with chronic WAD grades 2 and 3, will be recruited.

Intervention Group A, neck-specific exercises at a physiotherapy clinic: Participants get an explanation and justification for the exercise. They undergo a 12-week training program with a physiotherapist 2 times/week. Exercises are chosen from a clear and written frame of exercises, although the dosages are individually adapted. The training includes exercises activating the deep neck muscles, continuing with the endurance training of neck and shoulder muscles. The exercises are individually adjusted according to the individual's physical conditions and progressively increased in severity and dose. Exercise-related pain provocation is not accepted. The individual may also carry out home exercises. At the end of the treatment period, the patient is encouraged to continue practicing on their own.

Group B, neck-specific exercises with Internet support: Participants receive the same information and training programs as group A but have in total only four visits (a first examination visit and additional three visits) to the physiotherapist. When the exercises are introduced, they are repeated, and control is done so that the patient has understood how to conduct the exercises. The exercises take place, with the help of Internet support outside the health care system, probably mostly at home. Photos and videos of the exercises, information, and answers to frequently asked questions are available on the Internet (web-based system designed by the project leaders at the University). Patients can contact a physiotherapist if necessary, and can normally expect an answer within 3 days.

Any important harms or unintended effects in each group will be collected by the test leaders.

Sample size Sample size calculations in the study regarding group differences are calculated by a statistician (non-inferiority trial, an assumption that treatment B is not worse than A), and power is calculated by the software "G-POWER" and is based on the primary outcome measurements WAI and NDI. Regarding WAI, it is considered important that the participants improve from poor to moderate work ability, i.e., an average of 6 increments in a scale 7-47 (can also be classified into four groups: poor, moderate, good, and excellent). With a significance level of 5% and a power of 80%, seven people in each classification group are required. To get seven people in the "poor group" requires 60 people in total. To detect a clinically relevant improvement in NDI of 7%, 47 participants per group are needed on the basis of 80% power at a significance level of 5%. This value is based on the standard deviation (SD 13.4) in the NDI in a previous study on neck-specific exercises of individuals with chronic WAD grades 2 and 3. To ensure that enough people are in each group after drop-outs, for prediction analyses, and some possibility for subgroup analyses (e.g., WAD grades 2 and 3 or between men and women), the recommendation from the statistician was to include 70 people/group.

Ethical considerations The study was approved by the regional ethical review board (Linköping Dnr 2016 / 135-31). A previous clinical study relating to three different exercise interventions on long-term problems after whiplash injury demonstrated good efficacy of neck-specific exercise performed in primary health care. Current treatment is according to the best scientific evidence, and exercises used in the present study have been used in daily clinical practice for decades in the rehabilitation of various forms of neck pain. Participants are included after a thorough clinical examination and signed informed (oral and written information) consent. The exercises are adjusted individually. A risk of muscle soreness is present, but otherwise no negative side effects are to be expected.

Login is required to fill in Internet-based surveys and to gain access to the Internet-based exercise program. People with long-term problems often have low access to assessments and treatments as more acute conditions often are prioritized in the health care system. Both groups in the present study get active care that is expected to increase work ability. The benefit is deemed to be great, and there are no commercial interests.

The results will be presented at group level, and no connection to the individual person can be made. All data are anonymous and subject to the official health secrets act.

Statistical analysis Analyses will be done with parametric or non-parametric statistics, depending on the type of data and if the analysis is between groups or over time. Analyses will primarily be made on an intention-to-treat basis and as secondary as per protocol analysis. When suitable a linear mixed model analysis will be used. For prediction analysis, multivariate analysis will be performed. For calculation of cost-effectiveness, quality-adjusted life-years and incremental cost-effective ratios will be calculated.

Sub-group analyses regarding gender, WAD grade, neurology, headache, dizziness and compliance may be done.

Ultrasound registrations, electromyopgraphy, Magnetic Resonance Imaging and kinesthesia may be done on a sub-group of participants to investigate neck muscle structure and function. Interviews may be performed on a sub group of individuals to investigate the experience of function and study participation.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a whiplash injury in a traffic accident with a four-wheeled motor vehicle at least 6 months ago but less than 5 years ago, with chronic neck problems corresponding to Quebec Task Force (QTF) grades 2-3 verified in clinical examination
* No participation in a neck-specific exercise program in a previous research study;
* Average estimated pain in the preceding week more than 20 mm on the visual analogue scale (VAS)
* Neck disability for more than 20% of the Neck Disability Index
* Working age, between 18 and 63 years
* Daily access to computer/tablet/smart phone and Internet
* Time to follow the treatment program
* Neck symptoms within the first week after the injury (neck pain, neck stiffness, or radiculopathy from the neck).

Exclusion Criteria:

* Any of the following signs of brain damage at the time of injury: loss of consciousness, amnesia before or after the injury, altered mental status (e.g., confusion, disorientation), focal neurological changes (changes in smell and taste)
* Previous fractures or dislocation of the cervical column
* Known or suspected serious physical pathology included myelopathy, spinal tumours, spinal infection, or ongoing malignancy
* Previous severe neck problems that resulted in sick leave for more than a month in the year before the current whiplash injury
* Surgery in the cervical column
* Generalized or more dominant pain elsewhere in the body
* Other illness/injury that may prevent full participation in the study and/or where neck exercises are contraindicated
* Inability to understand and write in Swedish
* Diagnosed severe mental illness, e.g., psychosis, schizophrenia, personality disorders
* Current alcohol or drug abuse.

Ages: 18 Years to 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index (NDI) | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Self-reported neck-specific function

SECONDARY OUTCOMES:
Whiplash Disability Questionnaire | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Disability associated with whiplash
Patient-specific functional scale (PSFS) | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Individual ratings of function
Pain intensity in neck, head, and arm and dizziness by a VAS (0-100 mm) | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Pain intensity
Distribution of pain by a pain drawing assessed with images | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Distribution of pain
Frequency of pain | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Frequency of pain
Use of pain medications | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Use of pain medications
Dizziness/balance by the Dizziness Handicap Inventory (DHI) | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Dizziness questionnaire
Headache Questions by VAS and the Headache Impact Test (HIT-6) | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Impact of headache
Pain Catastrophizing Scale | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Self-reported pain catastrophizing
EuroQuol five dimensions | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Self-reported health
Effort Reward Imbalance questionnaire | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Work related balance between effort and reward
Symptoms Satisfaction scale | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Satisfaction with present symptoms
Physical activity score, a combination score of the 2 questions (everyday physical activity and exercise/sport/open-air activity) to a combined 4-point score | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Physical activity
Health care consumption, number of visits | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Health care consumption
Self-Efficacy Scale (SES) | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Self-reported self-efficacy
Fear Avoidance Beliefs Questionnaire (FABQ) | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Fear Avoidance Beliefs
Hospital Anxiety and Depression Scale | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Depression and anxiety
Post Traumatic Stress Disorder checklist (PCL-S) | Baseline
  Post Traumatic Stress
Range of neck motion | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Range of motion
Ergonomics questions and how work is perceived | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Work ergonomics
Sickness presence by the Stanford presenteeism scale | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Sickness presence at work
Patient Enablement Instrument (PEI) questionnaire | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Patient enablement
Consumption of analgesic drugs prescribed through the drug registry | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Consumption of analgesic drugs
Sick-leave registration, number of days and episodes | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Sick-leave
Cognitive failures questionnaire (CFQ) | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Cognitive function
Sensorimotor control of the neck muscles, mm Hg | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Sensorimotor control
Neck muscle endurance of ventral and dorsal neck muscles in seconds | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Neck muscle endurance
Balance measured in seconds, standing on one leg with eyes closed | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Balance
Neurology such as reflexes, sensibility, muscle weakness, Spurling´s test, neural tension test | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Neurology
Ultrasound registrations may be measured in a sub-group, deformation and deformation rate | Change from baseline to 3 months follow-up
  Neck muscle function
MRI may be measured in a sub-group. | Change from baseline to 3 months follow-up
  Neck muscle structure and maybe function

OTHER OUTCOMES:
Background data such as age and gender | Baseline
  Background data such as age, gender, living circumstances
Work Ability Index (WAI) | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Self-reported work ability
Global rating of change scale | Change from baseline to 3 months and 15 months follow-up, measured at follow-ups
  overall change because of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Anneli Peolsson, Professor, Principal Investigator — Dep. Medical and Health Sciences, Physiotherapy, Linköping University, Linköping, Sweden; Gunnel Peterson, PhD, Study Chair — Dep. Medical and Health Sciences, Physiotherapy, Linköping University, Linköping, Sweden; Maria Landén Ludvigsson, PhD, Study Chair — Dep. Medical and Health Sciences, Physiotherapy, Linköping University, Linköping, Sweden
Locations (1):
- Anneli Peolsson, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dalal K, Peterson G, Peolsson A. Health related quality of life (HRQOL) from the perspective of patients with chronic whiplash-associated disorders (WAD) in Sweden. BMC Musculoskelet Disord. 2025 Feb 14;26(1):154. doi: 10.1186/s12891-025-08397-2. PMID 39953445
- [Derived] Peolsson A, Wirqvist S, Kammerlind AS, Peterson G. Effectiveness of neck-specific exercises with and without internet-based support on dizziness/unsteadiness in chronic whiplash-associated disorders: Secondary analyses of a randomised controlled trial. PLoS One. 2024 Oct 7;19(10):e0311145. doi: 10.1371/journal.pone.0311145. eCollection 2024. PMID 39374216
- [Derived] Peolsson A, Nilsing Strid E, Peterson G. Novel Internet Support for Neck-Specific Rehabilitation Improves Work-Related Outcomes to the Same Extent as Extensive Visits to a Physiotherapy Clinic in Individuals with Chronic Whiplash-Associated Disorders: A Prospective Randomised Study. J Occup Rehabil. 2024 Dec;34(4):873-883. doi: 10.1007/s10926-024-10176-0. Epub 2024 Mar 25. PMID 38526764
- [Derived] Peterson G, Peolsson A. Efficacy of Neck-Specific Exercise With Internet Support Versus Neck-Specific Exercise at a Physiotherapy Clinic in Chronic Whiplash-Associated Disorders: Multicenter Randomized Controlled Noninferiority Trial. J Med Internet Res. 2023 Jun 20;25:e43888. doi: 10.2196/43888. PMID 37338972
- [Derived] Peolsson A, Landen Ludvigsson M, Peterson G. Neck-specific exercises with internet-based support compared to neck-specific exercises at a physiotherapy clinic for chronic whiplash-associated disorders: study protocol of a randomized controlled multicentre trial. BMC Musculoskelet Disord. 2017 Dec 12;18(1):524. doi: 10.1186/s12891-017-1853-1. PMID 29233141